CLINICAL TRIAL: NCT05520996
Title: Impact of Ostracism on Prospective Memory in ADHD Children With or Without Emotional Dysregulation/ Impact de l'Ostracisme Sur la mémoire Prospective Chez Des Enfants Atteint de TDA/H Avec ou Sans dysrégulation émotionnelle.
Brief Title: Impact of Ostracism on Prospective Memory in ADHD Children With or Without Emotional Dysregulation
Acronym: IOM-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/0224/OB
Record Dates: First submitted 2022-03-14; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm study (Experimental): Memory test performed before and after cyberball task
  Interventions: Behavioral: Cyberball

INTERVENTIONS:
Behavioral: Cyberball — Social exclusion or ostracism can be measured by the Cyberball 5 task. The principle of Cyberball is based on the creation of a situation of exclusion through a computerized task. During this task, the participant passes a ball to 2 other players controlled by Artificial Intelligence (AI). The ball-passing method of AI-controlled players is determined in advance in the computer program code. A series of ball passing is carried out with initially an equal passing between the three participants and then an exclusive passing between the players controlled by an artificial intelligence

SUMMARY:
Assess the effect of exposure to a situation of social exclusion or ostracism on the prospective memory of children with ADHD

ELIGIBILITY:
Inclusion Criteria:

* Child with attention deficit disorder with or without hyperactivity (ADHD) according to the following criteria: score greater than 27 on the ADHD-RS scale or score greater than 65 on the Conners scale, and after clinical staff discussion
* Social security
* non opposition of parents and children to the study

Exclusion Criteria:

* Subject presenting elements in favor of a depressive disorder according to a clinical evaluation and on an evaluation by the CBCL scale
* Minor and/or parents who do not understand French
* Person under legal protection, adult guardianship or curatorship.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
difference between prospective memory tests performed before and after cyberball task | At inlcusion
  Promacy test is a Memory test performed before and after Cyberball task

CONTACTS AND LOCATIONS:
Locations (1):
- CHU - Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No